CLINICAL TRIAL: NCT03998969
Title: Efficacy of DA-5204 (Stillen 2X®) for Patients With Gastroesophageal Reflux Disease: A Randomized, Double-blind, Placebo-controlled Pilot Study
Brief Title: Efficacy of DA-5204 on Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dong Ho Lee, Director, Clinical Research, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUBH-DHLDA5204
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Disease
Keywords: Gastroesophageal Reflux; Esophagitis, Peptic
MeSH Terms: conditions — Esophageal Diseases; Gastroesophageal Reflux; Esophagitis, Peptic | interventions — Pantoprazole; DA-5204

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pantoprazole and DA-5204 (Experimental): Pantoprazole 40mg once daily and 'DA-5204' twice daily by mouth, administered for 4 weeks
  Interventions: Drug: Pantoprazole; Drug: DA-5204
- Pantoprazole and placebo (Active Comparator): Pantoprazole 40mg once daily and 'placebo' twice daily by mouth, administered for 4 weeks
  Interventions: Drug: Pantoprazole; Drug: Placebo

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole 40mg tablet
  Other Names: Pantoline
Drug: DA-5204 — DA-5204 tablet
  Other Names: Stillen 2X®
  Arms: Pantoprazole and DA-5204
Drug: Placebo — Film-coated tablet manufactured to mimic DA-5204
  Other Names: Placebo (for DA-5204)
  Arms: Pantoprazole and placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled clinical Study to evaluate the efficacy of DA-5204 and proton pump inhibitor combination therapy compared with proton pump inhibitor alone therapy in patients with gastroesophageal reflux Disease.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a condition in which reflux of stomach contents into the esophagus causes troublesome symptoms, such as heartburn and acid regurgitation.

Proton pump inhibitors, as acid suppressor, are the agents recommended as the first-line treatment for gastroesophageal reflux disease. However, approximately 20-30% of patients have insufficient effect on this therapy alone.

DA-5204 is a medicine based on Artemisia asiatica 95% ethanol extract. DA-5204 has been administered to treat gastritis and gastric ulcers with antioxidative and cytoprotective actions on gastric mucosal damage. Therefore, we expect DA-5204 to be effective in reflux esophagitis (esophageal mucosal injury).

ELIGIBILITY:
Inclusion Criteria:

* Age is over 20 years old, under 75 years old, men or women
* Patients diagnosed with erosive esophagitis by gastroscopy
* Signed the informed consent forms

Exclusion Criteria:

* Patients who is impossible to receive gastroscopy
* Patients with esophageal stricture, esophageal varix, Barrett's esophagus, peptic ulcer or gastrointestinal bleeding
* Patients administered with prokinetics, H2 receptor antagonists, proton pump inhibitors, anticholinergic drugs or non-steroid anti-inflammatory drugs prior to study in 4 weeks
* Patients with surgery related to gastroesophageal
* Patients with Zollinger-Ellison syndrome
* Patients with any kind of malignant tumor
* Patients administered with anti-thrombotic drugs
* Patients with significant cardiovascular, pulmonary, heptic, renal, hemopoietic or endocrine system primary disease
* Patients with neuropsychiatric disorder, alcoholism, or drug abuse
* Patients taking other investigational drugs or participating in other clinical studies in 4 weeks.
* Women either pregnant or breast feeding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Endoscopically effective improvement | 4 weeks
  A percentage of subjects showed effective improvement of erosive esophagitis (esophageal mucosal injury) by the endoscopy.
  The definition of "effective improvement" is the subjects showed score changed from 3 to 0, from 2 to 0, or from 3 to 1.
  [score 0(LA grade N): normal mucosa, score 1(LA grade M): minimal changes to the mucosa such as erythema, blurring and/or whitish turbidity, score 2(LA grade A): non-confluent mucosal breaks <5 mm in length, score 3(LA grade B): non-confluent mucosal breaks ≥5 mm in length]
Endoscopically complete improvement | 4 weeks
  A percentage of subjects showed complete improvement of erosive esophagitis (esophageal mucosal injury) by the endoscopy.
  The definition of "complete improvement" is the subjects showed score changed from 3 to 0 or from 2 to 0.

SECONDARY OUTCOMES:
Symptom improvement | 4 weeks
  A percentage of subjects showed sufficient improvement of reflux symptom score from Gastroesophageal Reflux Disease Questionnaire (GerdQ).
  The definition of "sufficient improvement" is the subjects showed ≥50% reduction from the initial sum of scores for GerdQ.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bungdang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No